CLINICAL TRIAL: NCT00918437
Title: Characterization of the Postoperative Pain Course and Intensity After Uvulopalatoplasty With Radiofrequency Knife (RAUP)
Brief Title: Postoperative Pain Course After Uvulopalatoplasty
Status: Completed | Type: Observational
Sponsor: Ullevaal University Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Professor Lasse A. Skoglund, Section of Dental Pharmacology and Pharmacotherapy, University Of Oslo
Organization: Oslo University Hospital (Other)
Other Study IDs: OES-002
Record Dates: First submitted 2009-06-09; First posted 2009-06-11 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2005-06

CONDITIONS: Snoring; Surgical Procedures, Operative; Pain, Postoperative; Quality of Life
Keywords: uvulopalatoplasty; postoperative pain; quality of life
MeSH Terms: conditions — Snoring; Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- RAUP treatment: Patients referred to the hospital for a snoring problem

SUMMARY:
The aim of this study is to determine the postoperative course including effects on the quality of life following soft palate surgery with radiofrequency knife (RAUP).

DETAILED DESCRIPTION:
For the treatment of social snoring one common treatment modality is the surgical reconstruction of the soft palate. The procedure is a routine operation performed at nearly all Ear-Nose- and Throat departments in Norway. The surgery is done with local anaesthesia in an out-patient setting where the patients' postoperative observation at the hospital is limited to 1-2 hours. As the surgery is done in the sensitive mucosa and palatopharyngeal musculature the postoperative course might be unpleasant. The patients are therefore in the need of regular postoperative pain treatment extending into the 2 first weeks after surgery.

At hospitals the uvulopalatoplasty is performed using a radiofrequency knife (RAUP) after the soft palate has been infiltrated with local anaesthesia (1% xylocain/adrenaline). The incision is done paramedialy to the uvular base and up into the musculature of the soft palate then making a smooth arch toward the pharyngeal tonsil upper limit. The then elongated uvula is amputated to about ½ cm. Occasionally, a suture is placed laterally and medially to lift the palate and prevent postoperative scaring. Coagulation is done if necessary with light bipolar diathermy.

As the postoperative course might be unpleasant after RAUP it is of interest to study the time course and intensity of pain after surgery when using the standardised postoperative pain treatment at OmniaSykehuset. The result will be useful in future studies looking at ways to improve the pain treatment after uvulopalatoplasty.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex of Caucasian origin who are referred to the hospital for snoring that have been subjected to a sleep study indicating that uvulopalatoplasty might have a considerable affect on the snoring.

Exclusion Criteria:

* Chronic drug treatment (except birth control medication) with analgesics, anti-inflammatory treatment (both steroidal (SAIDs) and non-steroidal anti-inflammatory drugs (NSAIDs)) apart from standard postoperative analgesic treatment administered by the operator.
* Patients with diabetes.
* Patients who due to age or communication skills are considered unable to complete patient forms.
* Professional evaluation suggests an alteration of the planned surgical area or treatment form.
* Known or assumed intolerance or hyper sensibility to diclofenac, codeine or paracetamol (standard postoperative analgesic treatment).
* Consumption of alcohol in the period from 2 days before or until the end of the primary observation period (postoperative days 0-7

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of either sex, of Caucasian origin, between the age of 18 and 80, who are referred to the hospital for snoring that have been subjected to a sleep study indicating that uvulopalatoplasty might have a considerable affect on the snoring.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2005-06; Primary Completion 2008-05 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Pain Intensity 0-10 Numerical Rating Scale | 14 days

SECONDARY OUTCOMES:
Norwegian McGill Pain Questionnaire (NMPQ) | 14
Norwegian Translated Short-Form McGill Pain Questionnaire (NTSF-MPQ) | 14 days
Oral Health Impact Profile (OHIP-14) | 14 days
Corahs Dental Anxiety Scale (CDAS) | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Øystein S Eskeland, MD, Principal Investigator — University of Oslo; Lasse A Skoglund, DDS, DSci, Study Chair — University of Oslo; Per Skjelbred, MD, DDS, Study Director — Ullevaal University Hospital
Locations (1):
- Aleris Hospital, Oslo, Norway

REFERENCES:
- [Background] Melzack R. The McGill Pain Questionnaire: major properties and scoring methods. Pain. 1975 Sep;1(3):277-299. doi: 10.1016/0304-3959(75)90044-5. PMID 1235985
- [Background] Melzack R. The short-form McGill Pain Questionnaire. Pain. 1987 Aug;30(2):191-197. doi: 10.1016/0304-3959(87)91074-8. PMID 3670870
- [Background] Slade GD. Derivation and validation of a short-form oral health impact profile. Community Dent Oral Epidemiol. 1997 Aug;25(4):284-90. doi: 10.1111/j.1600-0528.1997.tb00941.x. PMID 9332805
- [Background] Corah NL. Dental anxiety. Assessment, reduction and increasing patient satisfaction. Dent Clin North Am. 1988 Oct;32(4):779-90. PMID 3053270
- [Background] Kim HS, Schwartz-Barcott D, Holter IM, Lorensen M. Developing a translation of the McGill pain questionnaire for cross-cultural comparison: an example from Norway. J Adv Nurs. 1995 Mar;21(3):421-6. doi: 10.1111/j.1365-2648.1995.tb02722.x. PMID 7745193